CLINICAL TRIAL: NCT06482346
Title: Clinical Pharmacology Study of MT-3534 in Healthy Adult Male Volunteers (SAD Study)
Brief Title: Clinical Pharmacology Study of MT-3534 in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MT-3534-Z-101; jRCT2031240187 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Healthy Adult Male Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MT-3534 (Experimental): Intravenous (IV)
  Interventions: Biological: MT-3534
- Placebo (Placebo Comparator): Intravenous (IV)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MT-3534 — Solution for infusion; Intravenous (IV)
  Arms: MT-3534
Biological: Placebo — Solution for infusion; Intravenous (IV)
  Arms: Placebo

SUMMARY:
This study is planned to investigate the safety, tolerability, and pharmacokinetics when a single intravenous dose of MT-3534 or a placebo is given to healthy adult male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male volunteer
* Japanese (Part A) or White (Part B)
* Subjects with age of 18 to 55 years old at informed consent
* Subjects with a full understanding of the nature of this study and consented in writing to participate in the study

Exclusion Criteria:

Additional screening criteria check may apply for qualification:

* Subjects with a current or prior disease history of cardiac, hepatic, renal, gastrointestinal, respiratory, neuropsychiatric, hematopoietic, endocrine systems, etc. whom the investigator has judged to be unfit for study participation
* Subjects with a history of drug or food allergies
* Subjects with a history of hypersensitivity to any of the ingredients of MT-3534
* Subjects whose BMI is less than 18.5 kg/m^2 or exceeds 25.0 kg/m^2, or subjects weighing less than 50.0 kg or exceeds 80.0 kg at the time of screening or Day -1 tests (Part A). Subjects whose BMI is less than 18.5 kg/m^2 or exceeds 30.0 kg/m^2, or subjects weighing less than 50.0 kg or exceeds 100.0 kg at the time of screening or Day -1 tests (Part B). (For BMI, values rounded to the first decimal place will be used.)
* Subjects who have donated blood or from whom blood samples have been collected in a total amount of 400 mL or more in the 12 weeks, 200 mL or more in the 4 weeks, or 800 mL or more in the 52 weeks prior to informed consent
* Subjects who have donated blood platelets or from whom blood samples have been collected in the 2 weeks prior to informed consent
* Subjects with a current or prior history of dependence on drugs, alcohol, etc
* Subjects with a history of cancer
* Subjects who receive a live attenuated vaccine within 4 weeks before the start of investigational product administration
* Subjects with a positive result for serological test for syphilis, Hepatitis C virus (HCV) antibody, or HIV antigen/antibody at screening
* Subjects with a positive result for Hepatitis B virus surface (HBs) antigen, Hepatitis B virus core (HBc) antibody and HBs antibody at screening (Subjects with a negative for HBs antigen plus a positive for HBs antibody plus a negative for HBc antibody and who have obvious history of vaccination are eligible to enroll)
* Subjects with a history of recurrent infections such as Herpes simplex or Herpes zoster
* Subjects with a positive result for polymerase chain reaction (PCR) test for COVID-19 at Day -1 test
* Subjects who do not agree to contraception from the date of informed consent until 12 weeks after the end of the administration of the investigational product
* Subjects who have participated in other clinical studies and received other investigational products within 12 weeks before informed consent
* Subjects who have used any drug other than the investigational product in the period within the 7 days before the start of investigational product administration or 5 times the half-life of the drug, whichever is longer
* Subjects judged by the investigator (or subinvestigator) to be ineligible for the study for any other reason

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to Day 85
Number of subjects with adverse reactions | up to Day 85
Serum concentrations of MT-3534 | up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Clinical Research Hospital Tokyo, Shinjuku-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No